CLINICAL TRIAL: NCT06409065
Title: Psycho-Spiritual Management for Patients With Advanced Cancer and Their Family Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-0450; NCI-2024-03804 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Attention Control (Experimental): Participants will take part in a meditation program. As part of this program, participants will complete up to 4 meditation sessions with a trained counselor. Participants should attend each session together as a family. All sessions will be online by videoconference using Zoom.
  Interventions: Behavioral: Meditation Program
- Behavioral Intervention (FFM Program) (Experimental): Participants will take part in a discussion program. Participants will be asked to complete 4 discussion sessions with a trained counselor over a course of a 4 week period. Participants should attend each session together as a family.
  Interventions: Behavioral: Meditation Program
- Usual Care (Experimental): All participants will receive cancer treatment per usual care (UC).
  Interventions: Behavioral: Meditation Program

INTERVENTIONS:
Behavioral: Meditation Program — Meditation and discussion sessions will be audio recorded
  Other Names: Discussion Program

SUMMARY:
The goal of this behavioral research study is to learn about the effects of two different supportive care programs on patients' and their family caregivers' psychological wellbeing and overall quality of life.

DETAILED DESCRIPTION:
To enhance the accessibility and scalability for future research, both the interventions (FFM and AC) will be delivered via videoconferencing. To increase the generalizability of the findings, a multi-site enrollment recruitment strategy will be used to enroll a diverse (including underserved) patient population. The program will be delivered in both English and Spanish and a varied social economic population will be enrolled in the program.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed with a metastatic (stage IV) breast, thoracic, gastrointestinal, gynecological, or genitourinary cancer
* Be without disease progression for at least 3 months based on surveillance CT imaging
* Have an ECOG performance status of ≤2
* Have a family caregiver willing to participate

Both patient and caregiver must meet all the following criteria:

* Be ≥18 years old
* Be able to read and speak English or Spanish.
* Be able to provide informed consent

Additionally, either the patient and/or caregiver must:

• Have a NCCN Distress Thermometer score of ≥4

Exclusion Criteria:

A patient who meets the following criteria will be excluded from participation in this study:

• Have cognitive deficits that would impede the completion of self-report instruments as deemed by their attending oncologist

3.3 Vulnerable Populations This study is designed for individuals who are at least 18 years of age, and there is no upper age limit. Children under the age of 18 will not be included. First and foremost, it is unlikely that a minor is diagnosed with a metastatic solid tumor. It is also unlikely that a minor serves as the primary family caregiver of a patient with cancer. Additionally, the intervention is designed for adults, and the assessment tools are not validated for minors. While pregnant caregivers (self-identified) are study eligible, we will also exclude pregnant patients (medical notes).

3.4 Recruitment/Screening Process Eligible study participants (i.e. cancer patients) will be identified using the electronic clinic appointment systems on their tumor characteristics (i.e. cancer type and stage) and date of birth (i.e. minimum 18 years old). Potential patients and caregivers will be approached during patients' appointment at an outpatient oncology appointment, screened for eligibility, and consented. Since this is a family-based intervention, it is possible that caregivers will not be present during the patients' clinic visits. If so, patients will be asked for permission to contact the caregiver via phone to obtain consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Depressive Symptoms | Through study completion; an average of 1 year.
  Participants will complete the Center for Epidemiologic Studies Depression Scale (CES-D), a 20-item self-report measure focusing on the affective component of depression, which is appropriate as patients may experience somatic symptoms due to treatment toxicities rather than depression.

CONTACTS AND LOCATIONS:
Overall Officials: Kathrin Milbury, MD,PHD, Principal Investigator — MD Anderson
Locations (1):
- MD Anderson, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2025-01-15): https://cdn.clinicaltrials.gov/large-docs/65/NCT06409065/ICF_000.pdf